CLINICAL TRIAL: NCT06520696
Title: Multi-modal Intervention for Lactation Care (MILC)
Brief Title: MILC: A Comprehensive Mobile Application That Addresses the Breastfeeding Challenges of Low-income Hispanic Mothers
Acronym: MILC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benten Technologies, Inc. (Industry)
Collaborators: RTI International (Other); Temple University (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); UConn Health (Other)
Responsible Party: Principal Investigator, Tony Ma, Project Director or Principal Investigator, Benten Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MILC; R44MD017174 (NIH)
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Breastfeeding, Exclusive
Keywords: breastfeeding; breastfeeding education; breastfeeding support; exclusive breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Eligible Hispanic participants in their third trimester will be recruited for the study. The intervention group will receive standard WIC services plus the MILC application. Participants will be asked to participate in the periodic follow-up assessments at 1, 3, and 6 months along with demonstrating breastfeeding via the MILC app. Participants in the control group will receive standard breastfeeding services from the WIC program and will be asked to participate in the periodic follow-up assessments at 1, 3, and 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: MILC application (Experimental): Eligible Hispanic participants in their third trimester will be recruited for the study. The intervention group will receive standard WIC services plus the MILC application.
  Interventions: Behavioral: MILC application
- Control Group: Usual Care (Experimental): Participants in the control group will receive care as usual with standard breastfeeding services from the WIC program.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: MILC application — Eligible Hispanic participants in their third trimester will be recruited for the study. Intervention group will receive standard WIC services plus the MILC application. Standard WIC support includes on-site lactation consultation, bilingual peer counseling, weekly peer support meetings, free breast pump, and enhanced food package for BF mothers. If a participant has trouble with breastfeeding, she will be referred to a home-visiting breastfeeding peer counselor in the area. Participants will be asked to participate in the periodic follow-up assessments at 1, 3 and 6 months along with demonstrating breastfeeding via MILC app. Participants will send in 1 BF video per month using the MILC app to verify continued BF and fill out monthly self-report to verify EBF. Participants in the incentive group will receive escalating monthly points as incentives for every additional month of continued BF and EBF.
  Arms: Intervention group: MILC application
Behavioral: Usual care — Participants in the control group will receive care as usual with standard breastfeeding services from the WIC program and will be asked to participate in the periodic follow-up assessments at 1, 3 and 6 months. Participants in the control group can receive financial compensation for the completion of assessments. This is necessary to maximize retention and adherence to the monthly assessment schedule, provide comparable remuneration as the incentive group, and minimize demoralization of control group participants following treatment assignment. All participants are informed of the differential group procedures during the randomization consent process. In addition to the follow-up assessment, control group will also complete a monthly self-report on BF status (both for EBF and "any BF"). For attention control purposes in this group, participants will be referred to a mobile app for tracking the baby's milestones called Baby Connect.
  Arms: Control Group: Usual Care

SUMMARY:
The innovative platform MILC is designed to provide an integrated and comprehensive professional and social support network with personalized breastfeeding (BF) education to target exclusive breastfeeding (EBF) and any BF behaviors in low-income Hispanic women. Formative research conducted for the development of MILC and results from pilot testing will help guide the completion of the development and testing of this prototype that specifically caters to Hispanic women. In the long term, MILC has the potential to increase the rates of EBF and any BF up to 12 months.

DETAILED DESCRIPTION:
Breastfeeding (BF) is positively associated with health benefits for infants. It reduces an infant's risks for various conditions such as respiratory tract infections, non-specific gastroenteritis, diarrhea, asthma, and sudden infant death syndrome (SIDS).

Despite high breastfeeding (BF) initiation of approximately 80% among the Hispanic population in the United States (US), less than 25% of infants were exclusively breastfed (EBF) through 6 months, further perpetuating ethnic disparities in chronic diseases such as diabetes, obesity, and hypertension. Hispanic women are more likely to supplement feeding with formula, than non-Hispanic or African American (AA) mothers. Research has reported that barriers such as insufficient BF education, lack of BF technical support (i.e. latching issues, sore nipples), returning to work, easy access to free or discounted formula milk from Women Infants and Children (WIC), lack of social support, perceived inconvenience, cultural belief that both formula and breastmilk (los-dos) is best for the babies, perception that the infant is not satiated, and embarrassment associated with breastfeeding result in premature weaning off BF among low-income Hispanic mothers. Therefore, increasing the duration of EBF and continuous BF among low-income Hispanic women would require an innovative and comprehensive approach that addresses the diverse range of barriers listed above.

The investigators hypothesize that MILC will show significantly higher percentages of BF mothers in the intervention group at each time (1 month, 3 months, and 6 months) point compared with the control group. In the short term, MILC will be shown to be usable and acceptable by Hispanic BF mothers to receive BF support, education, and guidance from primary care providers (PCP) and certified lactation consultants/international board certified lactation consultants (CLC/IBCLC). In the long term, the impact of MILC will increase the rates of EBF for up to 6 months along with increasing rates of any BF up to 12 months.

ELIGIBILITY:
Inclusion Criteria for focus groups:

* Mothers who successfully exclusively breastfed for up to 6 months, at least one child OR mothers who attempted EBF but were unsuccessful at breastfeeding, in the past 3 years
* Self-identify as Hispanic
* Be WIC-eligible
* Voluntarily consent
* Speak English

Inclusion Criteria for Randomized Control Trial (RCT):

* In their late third trimester (approximately 4 weeks from delivery)
* Can initiate BF immediately
* Self-identify as Hispanic
* Be WIC-eligible
* Voluntarily consent
* Not have psychiatric hospitalization within the last 3 months
* Not have current or suicidal thoughts or past attempts
* Own a smartphone device
* Speak English

Exclusion Criteria for focus groups and Randomized Control Trial (RCT):

1. Participants who are under the age of 18 or over 44
2. Women experiencing a fetal demise or infant death
3. Women who report the following conditions also will be excluded:

   * Human immunodeficiency virus (HIV)
   * Taking antiretroviral medication or chemotherapy agents
   * Untreated, active tuberculosis
   * T-Cell lymphotropic virus type I or type II
   * Illicit drug use
   * Receiving radiation therapy
   * Exposed to anthrax
   * Undergone breast surgery
   * Known exposure to environmental toxins
   * Active hepatitis B and C
   * Prescription drug use incompatible with lactation

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The proposed study seeks to enroll pregnant or post-partum Hispanic women. Given the focus of the proposed research, the study will only recruit female participants
Enrollment: 178 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Exclusive breastfeeding | 1 month, 3 months and 6 months
  Investigators will assess if participants are breastfeeding exclusively (EBF)through monthly self-reported information. Investigators will record information on EBF at 1 month, 3 months and 6 months among women in the intervention arm.
Any breastfeeding rate(EBF) | 1 month, 3 months and 6 months
  Investigators will assess if participants are continuous breastfeeding through monthly breastfeeding videos uploaded in the system. Investigators will report information on any breastfeeding at 1 month, 3 months and 6 months.

SECONDARY OUTCOMES:
Infant weight (Medical outcomes) | Baseline, 1 month, 3 months and 6 months
  Infant's weight using medical report collected at 1 month, 3 month and 6 months
Emergency department visit (Medical outcomes) | Baseline, 1 month, 3 months and 6 months
  Number of emergency department visited for infant will be collected at 1 month, 3 month and 6 months

OTHER OUTCOMES:
Latching | Baseline, 1 month, 3 months and 6 months
  It will be assessed using LATCH breastfeeding assessment scale. LATCH stands for latch, audible swallowing, type of nipple, comfort and hold. Each component is scored from 0-2. A LATCH score of 0-3 is regarded as poor, 4-7 as moderate, and 8-10 as good.
BF history & attitudes questionnaire | Baseline, 1 month, 3 months and 6 months
  New survey based on constructs that potentially moderate BF
Self-Efficacy Scale | Baseline, 1 month, 3 months and 6 months
  It will be assessed using the BF Self-Efficacy Scale Short Form (BSES-SF). The BSES-SF is a 14-item self-administered instrument derived from the original 33-item BSES that measures breastfeeding confidence. Total scores range from 14 to 70, with higher scores reflecting more significant levels of breastfeeding self-efficacy.
Iowa Infant Feeding Attitude | Baseline, 1 month, 3 months and 6 months
  It will be collected using the Iowa infant feeding attitudes scale (IIFAS). The scale is composed of 17 items for assessing attitude towards BF. The total IIFAS score can range from 17 to 85 with higher scores reflecting positive attitude towards breastfeeding
Acculturation | Baseline, 1 month, 3 months and 6 months
  It will be assessed by using the Acculturation Rating Scale for Mexican Americans II. The scale contains 48 items to which participants respond on a 5-point Likert scale ranging from "Not at all" to "Extremely often or almost always," with higher scores indicating greater cultural orientation.
Postnatal depression | Baseline, 1 month, 3 months and 6 months
  It will be assessed using Edinburgh Postnatal depression Scale (EPDS). The EPDS has a maximum score of 30; a score of 10 or more may indicate possible depression of varying severity.
Usability | Month 6 postpartum
  System Usability Scale (SUS)survey will be used to assess usability of the MILC app. A SUS score above 68 would be considered above average and anything below 68 is below average.
Acceptance and Adoption | Month 6 postpartum
  Technology Acceptance Model (TAM) will be used to assess acceptance of MILC app

CONTACTS AND LOCATIONS:
Overall Officials: Tony Ma, MS, Principal Investigator — Benten Technologies; Yukiko Washio, PhD, Principal Investigator — RTI International
Locations (3):
- United States (3):
  - UCONN Health, Farmington, Connecticut
  - RTI International, Research Triangle Park, North Carolina
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No